CLINICAL TRIAL: NCT00169923
Title: Anti-Inflammatory Effects of Rosiglitazone in Patients With Stage 4 and 5 Chronic Kidney Disease
Acronym: Hercules
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: it was not possible to recruit any patient in the study
Sponsor: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P06.108
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Kidney Disease; Inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
The purpose of this study in patients with stage 4 and 5 chronic kidney disease is to determine whether rosiglitazone can reduce inflammatory markers and to investigate its effect on intima media thickness, calcification and pulse wave velocity.

DETAILED DESCRIPTION:
This is a double-blind randomised placebo-controlled clinical multicenter trial in patients with stage 4 and 5 chronic kidney disease. Eligible patients in the outpatient kidney clinic and patients at the dialysis department will be informed by their treating physician about the study and they will be asked to join the study. Following informed consent the eligible patients will undergo baseline evaluation and will then be followed for a period of 48 weeks. Patients will be randomly divided in two groups: one group will take rosiglitazone (4 mg during the first 8 weeks once daily and 8 mg during the next 40 weeks once daily) and the other group will get placebo. The original medication will be continued. The total follow-up will be 48 weeks.

At the start of the study and at 4, 8, 12, 18, 24 and 48 weeks during follow-up inflammatory parameters (CRP, hs CRP, fetuin, fibrinogen), lipid profile,iron status, glucose and insulin will be measured. Intima media thickness, pulse wave velocity, bone densitometry,subjective global assessment will be performed at 0, 24 and 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Over 18 years of age
* Stage 4 or 5 chronic kidney disease according the K/DOQI guidelines

Exclusion Criteria:

* Life span of less than one year
* Alcohol abuse
* Transaminases > 2.5 times the upper limit
* Diabetes mellitus
* Pregnancy
* Cardiac disease with marked limitation of functional capacity (NYHA III or IV)
* Use of immunosuppressant agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
intima media thickness | 48 weeks

SECONDARY OUTCOMES:
carotid artery calcifications | 48 weeks
inflammation | 48 weeks
lipid profile | 48 weeks
metabolic profile | 48 weeks
pulse wave velocity | 48 weeks
nutritional status | 48 weeks
bone density | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: andré gaasbeek, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Medisch Centrum Haaglanden, The Hague, Z-Holland
  - Haga Ziekenhuis, The Hague, Z-Holland